CLINICAL TRIAL: NCT00476138
Title: Functional Effects of Epigallocatechingallate on Retinal Function in Glaucoma
Brief Title: Effect of Epigallocatechin-Gallate on Inner Retinal Function in Ocular Hypertension and Early Glaucoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: FISIONERVE-01
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Epigallocatechin-Gallate; Glaucoma; Optic Nerve; Pattern Electroretinogram; Retinal Ganglion Cells
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — epigallocatechin gallate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Epigallocatechin-gallate

SUMMARY:
The present study attempts to evaluate the potential beneficial effects of a flavonoid, the epigallocatechingallate, on retinal ganglion cell function, evaluated by pattern electroretinogram, in subjects with ocular hypertension or early glaucoma.

DETAILED DESCRIPTION:
Twenty ocular hypertension and twenty early open angle glaucoma patients will be randomly divided into two groups: 1. placebo group [ocular hypertension, n = 10, early glaucoma (n=10)], taking an oral placebo in addition to standard beta-blocker treatment for ocular hypertension; 2. Treatment group [ocular hypertension, n = 10, early glaucoma (n=10)], taking Epigallocatechingallate oral treatment (200 mg/day) in addition to standard beta-blocker treatment for ocular hypertension. The patients will undergo standard clinical examination including automated Humphrey perimetry (30-2), pattern electroretinogram recording and measurement of retinal nerve fiber layer thickness by Optical Coherence Tomography (OCT stratus) at baseline, 3 and 6 months of treatment and follow-up. All patients will be again tested at 3 and 6 months after changing, in a cross-over design, placebo with drug assumption and vice versa.

Main outcome measure will be pattern electroretinogram amplitude. Secondary measures will be Humphrey perimetry mean deviation and corrected pattern standard deviation, and the thickness of optic nerve fibers measured by OCT.

Pattern Electroretinogram recordings.

Stimuli will be horizontal gratings of 1.6 cycles/degree spatial frequency, modulated in counterphase at 8.14 Hz and electronically generated on a high-resolution TV monitor (contrast: 70%; mean luminance: 80 cd/m2; field size: 31° [width] x 24° [height]). Subjects fixate at the center of the stimulating field with natural pupils, whose size will be measured, at a viewing distance of 57 cm. The subjects or patients will wear full refractive correction for the test distance. Signals will be recorded by a standard, flat-cup, 9 mm Ag/AgCl electrode taped on the skin of the lower eyelid. A similar electrode, placed over the eyelid of the contralateral, unstimulated eye, will be used as reference. Responses will be amplified (100, 000), bandpass filtered (1-30 Hz), sampled with a resolution of 12 bits and averaged (250 events) with automatic artifact rejection. Two replications will be obtained for each record to verify reproducibility. Peak-to-peak amplitude (in microV) of the Fourier analyzed response 2nd harmonic will be measured.

Retinal Nerve Fiber Thickness by OCT

All patients will undergo OCT imaging (software version 4.0.1, Carl Zeiss Meditec Ophthalmic Systems Inc, Dublin, CA) of the peripapillary RNFL. The instrument will be properly aligned after the subjects are comfortably seated with their head and chin firmly positioned against the relative rests. The OCT lens will be adjusted for the patient's refractive error. The subject will be instructed to stare at the internal fixation target with the eye under examination, to enable the optic disc to come into the window and to be successively centered. The Z-offset and the polarization will be adjusted to optimize the axial interval to the OCT scan and to maximize the reflective signal, respectively. The scan protocol will be the fast RNFL thickness 3.4 (3 circular scans consecutively performed, each 3.46 mm in diameter, centered on the optic disc and averaged to form a mean baseline). All scans will be acquired five times per eye during the same day, with short breaks between measurements, under dark room conditions. Images with eye movements during scans, poor centration, poor focus, or a signal strength less than 7/10 were excluded. The mean of 3 separate RNFL measurements (256 A-scans each) with the best optic disc centration, reproducibility of the signal profiles and signal strength will be used. Retinal thickness will be measured with the location of the vitreoretinal interface and the retinal pigment epithelium defining the inner and outer boundaries of the retina, respectively. The boundaries of the RNFL will be defined by first determining the thickness of the neurosensory retina. The location of the posterior boundary of the RNFL will be determined by evaluating each A-scan for a threshold chosen to be 15 dB greater than the filtered maximum reflectivity of the adjacent retina. Various machine-generated parameters will be used for evaluation of RNFL thickness, including RNFL average thickness over the entire cylindrical section and average RNFL thickness in each quadrant (inferior, superior, temporal and nasal). Abnormal RNFL measurements using OCT will be defined as mean or quadrantic thickness values outside 95% normal limits, based on the instrument's normative age-matched database, that will be confirmed on at least three out of five repeat scans. The reference values obtained from the normal control group included in the study will be also considered. The average RNFL thickness, inferior RNFL thickness, and the superior RNFL thickness have been shown to be the best discriminators for glaucoma by the Stratus OCT. These three measures will be the RNFL parameters analyzed in our study. One author (DM) will perform all the image acquisitions.

ELIGIBILITY:
Inclusion Criteria:

* IOP > 21 mmHg at the time of diagnosis
* Response to ipotensive therapy
* No visible alterations of the optical nerve head (if OHT)
* Visual field: normal (if OHT), < -6dB at diagnosis (if POAG)
* Alterations in PERG
* Familiarity for glaucoma (if OHT)

Exclusion Criteria:

* Change of ipotensive therapy
* Ocular surgery
* Other ocular pathologies
* Smokers

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
PERG | six months

SECONDARY OUTCOMES:
IOP | six months
Optical Coherence Tomography measurements of retinal nerve fiber layer thickness | six months

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Falsini, MD, Principal Investigator — Chatolic University of Sacred Heart, Roma; Tommaso Salgarello, M.D., Principal Investigator — Catholic University, Italy; Dario Marangoni, M.D., Principal Investigator — Catholic University, Italy
Locations (1):
- Catholic University, Policlinico A. Gemelli (Hospital), Rome, Italy

REFERENCES:
- [Background] Salgarello T, Colotto A, Falsini B, Buzzonetti L, Cesari L, Iarossi G, Scullica L. Correlation of pattern electroretinogram with optic disc cup shape in ocular hypertension. Invest Ophthalmol Vis Sci. 1999 Aug;40(9):1989-97. PMID 10440253
- [Background] Colotto A, Falsini B, Salgarello T, Iarossi G, Galan ME, Scullica L. Photopic negative response of the human ERG: losses associated with glaucomatous damage. Invest Ophthalmol Vis Sci. 2000 Jul;41(8):2205-11. PMID 10892864
- [Derived] Falsini B, Marangoni D, Salgarello T, Stifano G, Montrone L, Di Landro S, Guccione L, Balestrazzi E, Colotto A. Effect of epigallocatechin-gallate on inner retinal function in ocular hypertension and glaucoma: a short-term study by pattern electroretinogram. Graefes Arch Clin Exp Ophthalmol. 2009 Sep;247(9):1223-33. doi: 10.1007/s00417-009-1064-z. Epub 2009 Mar 17. PMID 19290537